CLINICAL TRIAL: NCT06095856
Title: Evaluation of Masseter and Anterior Temporalis Muscles Activity After Using Different Methods to Locate Centric Relation in Healthy Adults: A Randomized Cross-Over Clinical Trial
Brief Title: Evaluation of Masseter and Anterior Temporalis Muscles Activity After Locating Centric Relation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Tarek Nofal, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1723
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Centric Occlusion - Centric Relation Discrepancy (Disorder)
Keywords: centric relation, temporomandibular joint stability

STUDY DESIGN:
Intervention Model Description: The trial will be a "Cross-Over" clinical trial, with a wash-out period of 24 hours between investigated interventions, to set superiority, using 3 randomized groups of participants, and an allocation ratio of 1:1:1.
Who Masked: Outcomes Assessor
Masking Description: Double blinded study:
  * Blinding of the operator is not applicable.
  * Blinding of the participants is not applicable.
  * Outcome assessors and biostatistician will be blinded. Participants' identity and their corresponding study group will be concealed by assigning an identification number to all lab communications, data files and reports for the transfer of data to and from assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lf-La-Ks (Experimental): On the first day, baseline muscle activity will be measured by the sEMG, then, the leaf gauge will be used till centric relation is located, then, muscle activity will be recorded once more. On the second day, baseline muscle activity will be measured by the sEMG, then, the Lucia jig will be used till centric relation is located, then, muscle activity will be recorded once more.
  On the third day, baseline muscle activity will be measured by the sEMG, then, the Kois deprogrammer will be used till centric relation is located, then, muscle activity will be recorded once more.
  Patient satisfaction questionnaire will be handed-out to the participants and filled-out at the end of the third day.
  Interventions: Device: Leaf Gauge; Device: Lucia Jig; Device: Kois Deprogrammer
- La-Ks-Lf (Experimental): On the first day, baseline muscle activity will be measured by the sEMG, then, the Lucia jig will be used till centric relation is located, then, muscle activity will be recorded once more. On the second day, baseline muscle activity will be measured by the sEMG, then, the Kois deprogrammer will be used till centric relation is located, then, muscle activity will be recorded once more. On the third day, baseline muscle activity will be measured by the sEMG, then, the leaf gauge will be used till centric relation is located, then, muscle activity will be recorded once more.
  Patient satisfaction questionnaire will be handed-out to the participants and filled-out at the end of the third day.
  Interventions: Device: Leaf Gauge; Device: Lucia Jig; Device: Kois Deprogrammer
- Ks-Lf-La (Experimental): On the first day, baseline muscle activity will be measured by the sEMG, then, the Koid deprogrammer will be used till centric relation is located, then, muscle activity will be recorded once more. On the second day, baseline muscle activity will be measured by the sEMG, then, the leaf gauge will be used till centric relation is located, then, muscle activity will be recorded once more. On the third day, baseline muscle activity will be measured by the sEMG, then, the Lucia jig will be used till centric relation is located, then, muscle activity will be recorded once more.
  Patient satisfaction questionnaire will be handed-out to the participants and filled-out at the end of the third day.
  Interventions: Device: Leaf Gauge; Device: Lucia Jig; Device: Kois Deprogrammer

INTERVENTIONS:
Device: Leaf Gauge — Occlusal device used to locate centric relation of the jaws
Device: Lucia Jig — Occlusal device used to locate centric relation of the jaws
Device: Kois Deprogrammer — Occlusal device used to locate centric relation of the jaws and deprogram jaw muscles

SUMMARY:
Statement of the Problem:

To create optimum maxillomandibular relationships, ease discomfort, and restore function, occlusal devices are used, therefore, these devices are of great importance in the field of prosthodontics.

Literature is scarce regarding the effect of various methods used in locating centric relation on muscle activity, in addition to which method is most accepted by the patients for whom centric relation is being located.

Null hypothesis:

There will be no difference in Masseter and Anterior Temporalis muscles activity and patient satisfaction after using the Leaf Gauge, The Lucia Jig and the Kois Deprogrammer.

DETAILED DESCRIPTION:
Research Question:

Which of the investigated methods will result in lower masseter and anterior temporalis muscles activity reading after locating centric relation in healthy adults, and will be more accepted by the patient?

Rationale for Carrying out the Trial: For the patient:

The results of the trial will identify the most effective and patient friendly method for locating a centric position, which instructions are easy to follow and apply. Furthermore, reaching a centric position, using one of the investigated methods, will help ensure orthopedic stability before, during and after the treatment process.

For the dentist:

The results of the trial will help the dentist decide on which is the most reliable, valid and least technique sensitive method to choose when facing clinical situations requiring occlusal analysis, recording the patient's CR, or occlusal equilibration.

Choice of Comparators:

The control for the proposed study is a negative control. sEMG readings will be recorded before (-ve control) and after using any of the investigated methods and locating centric relation. Comparison between the pre and post readings for each method used will allow for evaluation of efficacy and reliability for each of the investigated methods.

Another reason for using a negative control is that, among the methods currently in the literature, not a single one was labelled the gold standard, nor a consensus has been reached as to which method checks most of the requirements of the ideal device used to locate the centric relation. Each method still has its advantages, disadvantages and most importantly, indications and contraindications.

Aim of the Study:

The aim of the proposed study is to evaluate Masseter and Anterior Temporalis muscles activity after using different methods: the Leaf Gauge, the Lucia Jig and the Kois Deprogrammer to locate centric relation in healthy adults (Primary Outcome). Furthermore, the study aims to evaluate the patient satisfaction after using each of the investigated methods (Secondary Outcome).

PICOS:

Population: Healthy adults with no history of TMD. Interventions:

I1: The Leaf Gauge I2: The Lucia Jig I3: The Kois Deprogrammer Control: - (-ve Control)

Outcomes:

Primary (O1): Masseter and Anterior Temporalis muscles activity Secondary (O2): Patient satisfaction Study Design: Randomized cross-over clinical trial

Interventions:

Interventions will be carried out by the principal investigator.

Initial examination and primary impressions:

Full medical and dental history will be taken from the participants and TMJ examination will be done to ensure that the eligibility criteria will be met.

Intraoral scans for the upper and lower arch and the buccal bite will be done for each participant. Impressions will be sent to the lab for the fabrication of the Kois Deprogrammer.

For Group Lf-La-Ks:

On the first day, baseline muscle activity will be measured by the sEMG, then, the leaf gauge will be used till centric relation is located, then, muscle activity will be recorded once more. On the second day, baseline muscle activity will be measured by the sEMG, then, the Lucia jig will be used till centric relation is located, then, muscle activity will be recorded once more.

On the third day, baseline muscle activity will be measured by the sEMG, then, the Kois deprogrammer will be used till centric relation is located, then, muscle activity will be recorded once more.

Patient satisfaction questionnaire will be handed-out to the participants and filled-out at the end of the third day.

For Group La-Ks-Lf:

On the first day, baseline muscle activity will be measured by the sEMG, then, the Lucia jig will be used till centric relation is located, then, muscle activity will be recorded once more. On the second day, baseline muscle activity will be measured by the sEMG, then, the Kois deprogrammer will be used till centric relation is located, then, muscle activity will be recorded once more. On the third day, baseline muscle activity will be measured by the sEMG, then, the leaf gauge will be used till centric relation is located, then, muscle activity will be recorded once more.

Patient satisfaction questionnaire will be handed-out to the participants and filled-out at the end of the third day.

For Group Ks-Lf-La:

On the first day, baseline muscle activity will be measured by the sEMG, then, the Koid deprogrammer will be used till centric relation is located, then, muscle activity will be recorded once more. On the second day, baseline muscle activity will be measured by the sEMG, then, the leaf gauge will be used till centric relation is located, then, muscle activity will be recorded once more. On the third day, baseline muscle activity will be measured by the sEMG, then, the Lucia jig will be used till centric relation is located, then, muscle activity will be recorded once more.

Patient satisfaction questionnaire will be handed-out to the participants and filled-out at the end of the third day.

Sample Size:

Sample size was calculated using a previous study as reference. This study aimed to compare the muscle activity of masseter and anterior temporalis muscles after using different methods to achieve centric relation in normal subjects According to this study, the response of matched pairs is normally distributed with standard deviation 4.01. If the estimated difference in the mean response of matched pairs is 4.5, the minimally accepted sample size is 8, with probability (power) 0.8. The Type I error probability associated with this test is 0.05. Total sample size was increased to 10 per group (Total sample size will be 30 for all groups). Sample size was calculated by using PS Software.

Data collection methods Muscle activity reading before and after using the investigated devices to locate centric relation will be recorded and logged into a Microsoft Excel sheet. Telephone numbers of all patients included the study will be recorded as a part of the written consent. All patients will be given a phone call at least a day before they must show up for each procedure. Analysis will be performed on a per-protocol basis; participants who do not show-up will not be included in the analysis.

Data management:

All data will be entered and saved electronically. Patient files are to be stored in numerical order and stored in secured file. Data will be encrypted using a password. All data will be maintained after completion of the study.

Statistical methods:

Handling of numerical/quantitative variables: Numerical data will be explored for normality by checking the data distribution using Kolmogorov- Smirnov and Shapiro-Wilk tests. Data will be presented as mean & standard deviation. If data will be normally distributed comparison between 2 different groups will be performed by using Independent t-test, comparison between 2 related groups will be performed by using Paired t-test, while comparison between more than 2 groups will be performed by using One Way ANOVA test followed by Tukey's Post Hoc test for multiple comparisons. If data will be non- parametric data comparison between 2 different groups will be performed by using Mann- Whitney test, comparison between 2 related groups will be performed by using Wilcoxon Signed Rank test, while comparison between more than 2 groups will be performed by using Kruskal-Wallis test.

Handling of categorial / qualitative variables: Data will be presented as frequency and percentages. All comparisons will be performed by using Chi square test.

Monitoring No formal data monitoring committee will be needed since it is a study with known minimal risks.

Harms Patients will be inquired about any possible side effects after using any of the investigated methods. Any temporary or permanent adverse effect will be recorded and documented. Post-operative pain is a minor side effect that can be associated with prolonged mouth opening; it will be managed by non-steroidal anti-inflammatory drugs and muscle relaxants in case of unbearable pain.

Audit No formal auditing committee is available.

Research Ethics Approval:

This protocol and the template informed consent form were reviewed by the Ethics Committee of Scientific Research - Faculty of Dentistry - Cairo University, and approved on July 31st, 2023. Approval number 1723.

Protocol Amendments:

Any modifications to the protocol which may have an impact on the conduct of the study, potential benefit of the patient or may affect patient safety, including changes of study objectives, study design, sample sizes, study procedures, or significant administrative aspects will require a formal amendment to the protocol. Such amendment will be agreed upon by the Council of Fixed Prosthodontics Department.

Informed Consent:

Principal investigator will introduce the trial to patients and provide full explanation of its aim and benefits in plain language. Patients will then be able to have an informed discussion with the investigator. Investigator will obtain written consent from patients willing to participate in the trial. All consent forms will be translated into Arabic.

Confidentiality:

All study-related information will be stored securely. All participant information will be stored in locked cloud-based files. All reports, data collection, processes, and administrative forms will be identified by a coded ID [identification] number only to maintain participant confidentiality. All records that contain names or other personal identifiers will be stored separately from study records identified by code number. All local databases will be secured with password-protected access systems.

Declaration of Interest:

No Conflict of interest is currently present. If there will be any conflict of interest it will be declared.

Access to Data:

The principal investigator and the supervisors will be given access to the data sets. All data sets will be password protected. To ensure confidentiality, data dispersed to project team members will be blinded of any identifying participant information.

Post-trial Care:

All patients will be followed up for one week after the clinical trial is over.

Dissemination Policy:

* Study results will be published in an indexed journal (Scopus or Web of Science) as partial fulfillment of the requirements for PhD degree in Fixed Prosthodontics.
* Topics suggested for presentation or publication will be circulated to the authors.

Biological Specimens:

No biological specimens will be collected from the study participants in the proposed study.

Statement of Originality:

The work contained in this protocol has not been previously submitted for a degree or diplomat in any higher education institution.

ELIGIBILITY:
Inclusion Criteria:

* (20-50) years old.
* Medically free.
* Full set of dentition (excluding the third molar).

Exclusion Criteria:

* Patients with bone or joint diseases.
* Patients with TMD.
* Patients with anterior cross-bite.
* Patients with open bite (dental or skeletal). -Patients with teeth mobility.
* Patients with parafunctional habits.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle Activity | immediately after the intervention
  Surface electromyogram will be used to measure right and left Masseter and Anterior Temporalis muscles activity (MicroVolt)

SECONDARY OUTCOMES:
Satisfaction assessed by the Visual Analogue Scale | through study completion, an average of 1 month
  Will be measured using a Visual Analogue Scale (VAS), minimum value is 1 (completely unsatisfied) and maximum value is 10 (completely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Amina A. Zaki, BDS,MSc,PhD, Study Chair — Cairo University; Reham S. Elbasty, BDS,MSc,PhD, Study Chair — Cairo University; John C. Kois, DMD,MSD, Study Chair — University of Washington
Locations (1):
- Faculty of Dentistry - Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carr AB, Donegan SJ, Christensen LV, Ziebert GJ. An electrognathographic study of aspects of 'deprogramming' of human jaw muscles. J Oral Rehabil. 1991 Mar;18(2):143-8. doi: 10.1111/j.1365-2842.1991.tb00041.x. PMID 2037936
- [Background] Hassall D. Centric relation and increasing the occlusal vertical dimension: concepts and clinical techniques - part one. Br Dent J. 2021 Jan;230(1):17-22. doi: 10.1038/s41415-020-2502-x. Epub 2021 Jan 8. PMID 33420450
- [Background] Hassall D. Centric relation and increasing the occlusal vertical dimension: concepts and clinical techniques - part two. Br Dent J. 2021 Jan;230(2):83-89. doi: 10.1038/s41415-020-2593-4. Epub 2021 Jan 22. PMID 33483662
- [Background] Adamczyk, Ł. and Więckiewicz, M. (2017) 'Clinical aspects of application of selected anterior deprogrammers', Protetyka Stomatologiczna, 67(4), pp. 333-341. doi: 10.5604/01.3001.0010.6860.
- [Background] Alqutaibi, A. Y. and Aboalrejal, A. N. (2015) 'Types of Occlusal Splint in Management of Temporomandibular Disorders (TMD)', Journal of Arthritis, 04(04). doi: 10.4172/2167-7921.1000176.
- [Background] Derwich M, Pawlowska E. Do the Mandibular Condyles Change Their Positions within Glenoid Fossae after Occlusal Splint Therapy Combined with Physiotherapy in Patients Diagnosed with Temporomandibular Joint Disorders? A Prospective Case Control Study. J Pers Med. 2022 Feb 10;12(2):254. doi: 10.3390/jpm12020254. PMID 35207741
- [Background] Gaikwad, A. M., Nadgere, J. and Tamore, S. (2022) 'Effect of muscle deprogrammers on muscle activity of masseter and temporalis muscles using surface electromyography: A randomized crossover clinical study', Journal of International Oral Health, 14(1), pp. 26-33. doi: 10.4103/JIOH.JIOH_208_21.
- [Background] Jayne, D. (2006) 'A deprogrammer for occlusal analysis and simplified accurate case mounting', Journal of Cosmetic Dentistry, 21(4), pp. 96-102.
- [Background] Land MF, Peregrina A. Anterior deprogramming device fabrication using a thermoplastic material. J Prosthet Dent. 2003 Dec;90(6):608-10. doi: 10.1016/j.prosdent.2003.09.011. PMID 14668765
- [Background] Lee DJ, Wiens JP, Ference J, Donatelli D, Smith RM, Dye BD, Obrez A, Lang LA. Assessment of occlusion curriculum in predoctoral dental education: report from ACP Task Force on Occlusion Education. J Prosthodont. 2012 Oct;21(7):578-87. doi: 10.1111/j.1532-849X.2012.00876.x. PMID 23130597
- [Background] Lucia, V. O. (1964) 'A Technique for Recording Centric Relation', Journal of Prosthetic Dentistry, 14(3), pp. 492-505.
- [Background] Machado NA, Henriques JC, Lelis ER, Tavares M, Almeida Gde A, Fernandes Neto AJ. Identification of occlusal prematurity by clinical examination and cone-beam computed tomography. Braz Dent J. 2013;24(1):64-7. doi: 10.1590/0103-6440201301974. PMID 23657416
- [Background] Sribabu, E. and Behera, S. S. P. (2018) 'Conceptions and misconceptions about centric relation: A Review of Literature', International Journal of Preventive and Clinical Dental Research, 5(2), pp. 44-48.
- [Background] Wiens JP, Goldstein GR, Andrawis M, Choi M, Priebe JW. Defining centric relation. J Prosthet Dent. 2018 Jul;120(1):114-122. doi: 10.1016/j.prosdent.2017.10.008. Epub 2018 Mar 8. PMID 29526300
- [Background] Wiens JP, Priebe JW. Occlusal stability. Dent Clin North Am. 2014 Jan;58(1):19-43. doi: 10.1016/j.cden.2013.09.014. PMID 24286644
- [Background] Zonnenberg AJ, Mulder J, Sulkers HR, Cabri R. Reliability of a measuring-procedure to locate a muscle-determined centric relation position. Eur J Prosthodont Restor Dent. 2004 Sep;12(3):125-8. PMID 15521396
- [Background] Zuccolotto MC, Vitti M, Nobilo KA, Regalo SC, Siessere S, Bataglion C. Electromyographic evaluation of masseter and anterior temporalis muscles in rest position of edentulous patients with temporomandibular disorders, before and after using complete dentures with sliding plates. Gerodontology. 2007 Jun;24(2):105-10. doi: 10.1111/j.1741-2358.2007.00152.x. PMID 17518958
- [Derived] Nofal AT, Kois JC, Elbasty RS, Zaki AA. Anterior temporalis and masseter muscle activity with different centric relation locating methods: A randomized cross-over trial. Sci Rep. 2025 Oct 13;15(1):35568. doi: 10.1038/s41598-025-21616-z. PMID 41083874